CLINICAL TRIAL: NCT06708364
Title: Effects of Virtual Reality Training on Heart Rate Variability and Recovery Heart Rate in Sedentary Individuals
Brief Title: Virtual Reality Training for Heart Rate Variability and Recovery Heart Rate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Rec/01894 Javeria Shahzadi
Record Dates: First submitted 2024-11-25; First posted 2024-11-27 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Sedentary Behavior
Keywords: Heart rate variability; Recovery Heart rate; Virtual Reality Training; Sedentary life style
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality Training (Experimental): Virtual reality training (X-BOX) for 6 weeks
  Interventions: Other: Virtual Reality Training
- Cycle Ergometer (Active Comparator): Aerobic activity on cycle ergometer for 6 weeks
  Interventions: Other: Cycle Ergometer

INTERVENTIONS:
Other: Virtual Reality Training — Virtual reality training (X-BOX). Table tennis
  * Frequency: 3 day per week
  * Intensity: Mild to moderate as per Game. Exer-game ( River Rush)
  * Time: total 30 minute of training with 5 min warm and 5 min cool down.
  * Type: aerobic exercise
  Arms: Virtual Reality Training
Other: Cycle Ergometer — * Frequency: 3 days per week.
  * Intensity: 40-60% of HRR
  * Time: total 30 minutes with 5 min warm up and 5 min cool down
  * Type: aerobic exercise
  Arms: Cycle Ergometer

SUMMARY:
To determine effects of VR training on Heart Rate Variability (HRV), Recovery Heart rate (RHR), Rate Pressure Product (RPP) and Rate of Perceived Exertion (RPE) in sedentary Individuals. Sedentary behavior is a significant public health concern associated with various chronic diseases and reduced quality of life. By elucidating the potential of virtual reality training as an innovative approach to promote physical activity and improve cardiovascular health, this research contributes to addressing the growing burden of sedentary lifestyle-related health conditions.

DETAILED DESCRIPTION:
Virtual reality (VR) training in cardiopulmonary rehabilitation (CR) offers an innovative approach to traditional exercise programs by incorporating enjoyable activities. Utilizing VR enhances cardiopulmonary endurance training and promotes the beneficial effects of CR by engaging patients in fun and challenging activities. This approach aims to increase motivation and adherence to CR over an extended period, resulting in improved mental and physical outcomes compared to conventional CR programs

ELIGIBILITY:
Inclusion Criteria:

* Sedentary Individuals (IPAQ-short version) < 3.3 METS daily
* Daily sitting time≤7 hours

Exclusion Criteria:

* Decline Consent
* Known cases of systemic or Cardiovascular Diseases.
* Obese (Asian BMI) > 29.9
* Any contra-indication to exercise/ Pregnancy

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2024-11-20 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-05-15 (Actual)

PRIMARY OUTCOMES:
Heart Rate Variability (HRV) | 2 weeks, 4 weeks, 6 weeks
  From baseline till 2nd, 4th, and 6th weeks measured through wireless ECG device which measures inter-beat (RR) intervals while doing physical activities. In adults , average HRV is 42 milliseconds.
Recovery Heart Rate | 2 weeks, 4 weeks, 6 weeks
  From baseline till 2nd, 4th, and 6th weeks measured through pulse oximeter. One-minute HRR for the average person is between 15 to 25 bpm, with a higher number indicating a quicker recovery and a potentially healthier heart.
Rate Pressure Product | 2 weeks, 4 weeks, 6 weeks
  Changes from baseline to 2 weeks, 4 weeks and 6 weeks after the intervention, measured through product of heart rate and systolic blood pressure, is a very reliable indicator of myocardial oxygen demand. An RPP above 20,000 mmHg per minute is considered healthy, whereas anything below 16,000 mmHg is considered insufficient.
Rating of Perceived Exertion (RPE) | 2 weeks, 4 weeks, 6 weeks
  Changes from baseline to 2 weeks, 4 weeks and 6 weeks after the intervention, measured through Borg RPE scale for measuring an individual's effort and exertion, breathlessness and fatigue during physical work. The RPE scale ranges from 6 to 20, each gradually related to the respondent's perceived exertion level.

CONTACTS AND LOCATIONS:
Overall Officials: Mehwish Waseem, MSPT-CPPT, Principal Investigator — Riphah International University
Locations (1):
- Pakistan Railway General Hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No